CLINICAL TRIAL: NCT03531177
Title: Healthy Eating & Active Lifestyle for Diabetes in UK African & Caribbean Communities: a Feasibility Trial With Process Evaluation
Brief Title: Healthy Eating & Active Lifestyles for Diabetes: Feasibility Trial
Acronym: HEAL-D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HEAL-DV2
Record Dates: First submitted 2018-05-03; First posted 2018-05-21 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Type2 Diabetes
Keywords: type 2 diabetes; Ethnicity; African-caribbean; Education; Self-management
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Randomised model, two arms. Intervention assessed against control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): HEAL-D diet and lifestyle education and behavioural change intervention, 7 sessions over 14 weeks.
  Interventions: Behavioral: HEAL-D
- Control (Active Comparator): Usual care.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: HEAL-D — HEAL-D is a 7 session programme of self-management education and behaviour change support for African and Caribbean patients with type 2 diabetes. The sessions will support participants with behaviour change to adopt evidence-based diet and physical activity targets for type 2 diabetes. The intervention has been systematically developed with defined theory and behavioural change techniques mapped to this theory.
  Arms: Intervention
Behavioral: Control — Participants receive usual care from their healthcare team.
  Arms: Control

SUMMARY:
The HEAL-D feasibility trial is a randomised control study to determine the feasibility of conducting an effectiveness trial of the Healthy Eating & Active Lifestyles for Diabetes programme; a culturally-tailored diet and lifestyle intervention for the management of type 2 diabetes in African and Caribbean communities. In this feasibility study HEAL-D will be evaluated against usual care in 80 patients with type 2 diabetes. HEAL-D is a programme of culturally-tailored diabetes self-management education and support, delivered over 7 sessions. Key outcomes are the acceptability of the programme; and recruitment and retention of the research participants. The current study will also pilot the feasibility and acceptability to participants of measuring proposed primary and secondary outcomes including HbA1c, blood lipids (triglyceride, total cholesterol, HDL-cholesterol, LDL-cholesterol), body weight, waist circumference, diabetes knowledge, diabetes and dietary competence, diabetes empowerment, perceived social support, quality of life, dietary intake, and physical activity.

DETAILED DESCRIPTION:
This study is a feasibility trial with an embedded process evaluation of the HEAL-D intervention compared with usual care. The study will use a randomised controlled trial (RCT) design, with individual patients as the unit of randomisation, evaluating the HEAL-D programme against usual care. The RCT design has been chosen primarily to evaluate the feasibility of recruiting and retaining a control arm, as well as to define what constitutes 'usual care' and the variability within that. Patients with diagnosed type 2 diabetes (T2D) will be recruited from General Practice surgeries in the London Boroughs of Lambeth and Southwark. In addition participants from the phase 1 co-design study will be invited to participate and self-referral methods will also be used, for example posters and advertisements in community locations. Patients will be eligible if they have a documented diagnosis of T2D and are of self-declared African or Caribbean ethnicity. Patients with complex therapeutic dietary needs may be ineligible if their individual needs are deemed incompatible with the aims of the intervention. Additionally patients who are unable to communicate in English will be ineligible.

A pragmatic sample size of 80 randomised patients, 40 in each arm, is anticipated to be sufficient to evaluate the programme, allowing for 20% drop-out/non-completion. As this is a feasibility trial it is not powered to detect statistically significant intervention effects, unless these estimated effects are extremely large. The purpose of the study is to assess the feasibility and acceptability of the intervention and of trial methods, and to provide estimates of key parameters such as potential effect sizes, recruitment and retention rates of the trial and participation rates of the programme, so that the optimal design of a full-scale trial can be determined.

The HEAL-D intervention consists of 7 sessions; the programme will have a flexible schedule allowing participants to attend either fortnightly or monthly sessions. Each patient who participates will be in the study for approximately 7 months and will be asked to complete two assessment visits, one at baseline and one 6-8 months later, depending on the intensity of programme attendance. A range of potential primary and secondary outcome data will be collected including HbA1c, blood lipids (triglyceride, total cholesterol, HDL-cholesterol, LDL-cholesterol), body weight, waist circumference, diabetes knowledge, diabetes and dietary competence, diabetes empowerment, perceived social support, quality of life, dietary intake, and physical activity. Participants may also participate in an interview or focus group as part of the study's process evaluation.

ELIGIBILITY:
Inclusion Criteria:

* documented diagnosis of type 2 diabetes
* self-declared African, Caribbean or Black British ethnicity

Exclusion Criteria:

* Complex dietetic needs e.g. advanced renal disease, making them unsuitable for general diet and lifestyle advice.
* Complex educational needs making them unsuitable for general group education.
* Unable to communicate in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2018-04-26 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
HbA1c | 6 months
  glycosylated hemoglobin, mmol/mol
Waist circumference | 6 months
  Waist circumference, cm

SECONDARY OUTCOMES:
Body weight | 6 months
  Body weight, kg
Total cholesterol | 6 months
  Total cholesterol, mmol/l
LDL-cholesterol | 6 months
  LDL-cholesterol, mmol/l
HDL-cholesterol | 6 months
  HDL-cholesterol, mmol/l
triglycerides | 6 months
  triglycerides, mmol/l
Diabetes knowledge | 6 months
  Measured using the Short Diabetes Knowledge Instrument
Perceived Diabetes & Dietary Competence | 6 months
  Measured using the Perceived Diabetes & Dietary Competence (PDDC) questionnaire
Diabetes Empowerment | 6 months
  Measured using the Diabetes Empowerment Scale-Short Form (DES-SF). It measures an individuals psychosocial self-efficacy with regard to their type 2 diabetes management. It uses a 5 point scale: Strongly Disagree; Somewhat disagree; Neutral; Somewhat Agree; Strongly Agree Strongly Disagree has a score of 1 through to strongly agree with a score of 5. The questionnaire is scored by averaging scores for all completed items. Total score ranges from a minimum of 1 to a maximum score of 5. The higher the score the higher the self-efficacy/empowerment. There are no sub-scales in this measure.
Perceived social support | 6 months
  Measured using the Multidimensional Scale of Perceived Social Support (PSS). It measures the degree to which an individual feels socially supported. Scores are on a numerical scale from 1 to 7 with 1 being the lowest social support and 7 the highest. The scores are summed. Three subscales are reported: family; friends; and significant other. Each subscale scores a minimum 4 and maximum 28. The total score ranges from 12 to 84.Higher scores indicate higher the degree of perceived social support.
Quality of Life | 6 months
  The EuroQol Five Dimension Three Level (EQ-5D-3L) scale measures health status. Level 1: respondents choose one statement which best describes their health status (5 dimensions: mobility, self-care, usual activities,pain/discomfort, and anxiety/depression), coded as 1 (no problems), 2 (some problems), or 3 (extreme problems). Numerals 1-3 have no arithmetic properties and should not be used as a cardinal score.The person's health status is defined by a 5-digit number, ranging from 11111 (no problems in all dimensions) to 33333 (extreme problems in all dimensions). There are potentially 243 different scores. Level 2 is the Visual Analogue Scale giving a score from 0 to 100, higher values indicating better health. The total score ranges from 0-1, it is calculated by applying a formula that essentially attaches values ('weights') to each of the levels in each dimension. The index can be calculated by deducting the appropriate weights from 1, the value for full health (i.e. state 11111).
Diabetes-specific Quality of Life | 6 months
  Measured using the Problem Areas In Diabetes-5 point scale (PAID-5). Each question has five possible answers with a value from 0 to 4, with 0 representing "no problem" and 4 "a serious problem". The scores for each of the 5 questions are added up to give a total score ranging from 0 to 20, with higher scores indicating higher degree of problems with diabetes.
Dietary carbohydrate intake | 6 months
  Measured in grams/day from a 24 hour recall interview
Physical activity | 6 months
  Measured as minutes of moderate intensity exercise per day using the Motion Watch accelerometer

CONTACTS AND LOCATIONS:
Overall Officials: Louise M Goff, PhD, Study Chair — King's College London; Barbara McGowan, PhD, Principal Investigator — Guy's and St Thomas NHS Foundation Trust
Locations (1):
- Guys and St Thomas NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moore AP, Rivas C, Harding S, Goff LM. A qualitative evaluation of the effectiveness of behaviour change techniques used in the Healthy Eating and Active Lifestyles for Diabetes (HEAL-D) intervention. BMC Public Health. 2025 Feb 11;25(1):568. doi: 10.1186/s12889-025-21767-8. PMID 39934762
- [Derived] Goff LM, Rivas C, Moore A, Beckley-Hoelscher N, Reid F, Harding S. Healthy Eating and Active Lifestyles for Diabetes (HEAL-D), a culturally tailored self-management education and support program for type 2 diabetes in black-British adults: a randomized controlled feasibility trial. BMJ Open Diabetes Res Care. 2021 Sep;9(1):e002438. doi: 10.1136/bmjdrc-2021-002438. PMID 34518159
- [Derived] Goff LM, Moore AP, Rivas C, Harding S. Healthy Eating and Active Lifestyles for Diabetes (HEAL-D): study protocol for the design and feasibility trial, with process evaluation, of a culturally tailored diabetes self-management programme for African-Caribbean communities. BMJ Open. 2019 Mar 1;9(2):e023733. doi: 10.1136/bmjopen-2018-023733. PMID 30826792